CLINICAL TRIAL: NCT00824707
Title: A Randomized, Controlled Study to Evaluate the Efficacy and Significant of the Anti-virus Therapy for the Unresectable Hepatitis B Virus-related Primary Liver Cancer
Brief Title: Efficacy and Significance of Antiviral Therapy for Unresectable Hepatitis B Virus-related Primary Liver Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBH-RCT-2008-005
Record Dates: First submitted 2009-01-16; First posted 2009-01-19 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Primary Liver Cancer
Keywords: primary liver cancer; hepatitis B virus; anti-virus therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B | interventions — entecavir; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- anti-virus therapy (Experimental): 100 HCC patients will be allocated to receive anti-virus therapy.
  Interventions: Drug: Entecavir
- conventional therapy (Active Comparator): 100 patients will undergo conventional therapy
  Interventions: Drug: conventional therapy

INTERVENTIONS:
Drug: Entecavir — Entecavir 0.5mg per day
  Other Names: anti-virus group
  Arms: anti-virus therapy
Drug: conventional therapy — conventional therapy including protecting the liver function, anti-tumor and so on
  Other Names: control group
  Arms: conventional therapy

SUMMARY:
This study is working to research the efficacy and significant of the anti-virus therapy in the unresectable Hepatitis B virus (HBV) related primary liver cancer(PLC) so as to establish treatment standards of anti-virus therapy in PLC.

DETAILED DESCRIPTION:
primary liver cancer(PLC)is one of the world's most common malignancies, especially in East-Asian countries.Hepatitis B virus (HBV) infection is associated with 70-90% of PLC cases in China. PLC can develop during any stage of the natural course of chronic HBV infection and anti-virus therapy should be considered during the management of PLC. However, there is no definite guide on when or how to practice the anti-virus therapy, especially in unresectable or inoperable PLC. Because of these facts, research on the significant of the anti-virus therapy in the HBV-related PLC is urgently needed.

200 patients will be randomly assigned to anti-virus therapy group and control gruop.The time to progression(TTP) and overall survival within two years will be used to evaluate the effect of anti-virus therapy on PLC.

The aim of this study is to research the efficacy and significant of the anti-virus therapy in the unresectable HBV-related PLC so as to establish treatment standards of anti-virus therapy in PLC.

ELIGIBILITY:
Inclusion Criteria:

1. Identify patients with PLC in accordance with the clinical diagnostic criteria of PLC.Patients with PLC shall be diagnosed with or without pathology. It is not appropriate to perform liver resection operation.
2. serum positive HBsAg≥6 months.
3. Criteria of liver function: Child A or B level, serum total bilirubin ≤ 1.5 times the upper limit of normal value, alanine aminotransferase and aspartate aminotransferase ≤ 10 times the upper limit of normal value.
4. hemoglobin≥8.5g/dl, PT-INR≤2.3 or PT>6 seconds of normal value.
5. No dysfunction in major organs; Blood routine, kidney function, cardiac function and lung function are basically normal.
6. Patients who can understand this trial, male or female, aged 18-70 voluntarily participate in clinical trials and have signed information consent.

Exclusion Criteria:

1. Patients with apparent cardiac, pulmonary, cerebric and renal dysfunction, which may affect the treatment of liver cancer.
2. Patients with other diseases which may affect the treatment mentioned here.
3. Patients with medical history of other malignant tumors.
4. Subjects participating in other clinical trials.
5. Women in pregnancy and breast-feeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2008-12; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
time-to-progression(TTP) | 1,2 and 3 years

SECONDARY OUTCOMES:
Overall survival (OS) | 1,2 and 3 years
The overall response rate | 1,2 and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shen Feng, M.D, Study Chair — Eastern Hepatobiliary Surgery Hospital
Locations (1):
- Eastern Hepatobiliary Surgery Hospital, Shanghai, Shanghai Municipality, China